CLINICAL TRIAL: NCT04588233
Title: Understanding the Impact of Melatonin Use on Adolescent Functioning: A Pilot and Feasibility Trial of the Melatonin Adolescent Research Study (MARS)
Brief Title: Melatonin Adolescent Research Study
Acronym: MARS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 5200334
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Sleep Disorders in Children
Keywords: Melatonin; Sleep Disturbance; Adolescents; Daytime Functioning
MeSH Terms: conditions — Parasomnias | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Administration of Melatonin (Experimental)
  Interventions: Dietary Supplement: Melatonin
- Administration of Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Each subject will receive 3mg of melatonin 1 hour prior to bedtime for 12 consecutive nights
  Arms: Administration of Melatonin
Other: Placebo — Each subject will receive a placebo 1 hour prior to bedtime for 12 consecutive nights
  Arms: Administration of Placebo

SUMMARY:
The present study will use a within-person, randomized cross-over experimental design to test the effects of exogenous melatonin supplementation on the sleep and daytime functioning of typically developing adolescents with short or disrupted sleep of behavioral origins (i.e., difficulty falling asleep, staying asleep, or premature waking resulting in short or disrupted sleep not attributed to an organic sleep condition).

ELIGIBILITY:
Inclusion Criteria:

* Self-identified sleep difficulties (e.g., difficulty falling asleep, staying asleep, or premature waking resulting in short or disrupted sleep).
* Ages 13 to 17 years old
* Able to understand, read, and write in English
* Melatonin naive

Exclusion Criteria:

* Obesity
* Use of psychiatric medication
* Drug(s), or supplements known to affect sleep
* History of head injury or concussion with loss of consciousness >1 minute
* Daily consumption of >1 caffeinated beverage
* Risk for any organic sleep disorder (e.g., obstructive sleep apnea, restless leg syndrome)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Objective Sleep Duration During Melatonin Administration | Change between baseline and two weeks
  Objective sleep will be measured via wrist-worn actigraphy worn nightly for 2 "run-in" nights followed by 12 consecutive nights after receiving melatonin (14 nights/2 weeks total). Changes in objective sleep duration would be demonstrated by either an increase or decrease in number of hours asleep compared to baseline
Change in Objective Sleep Duration During Placebo Administration | Change between baseline and two weeks
  Objective sleep will be measured via wrist-worn actigraphy worn nightly for 2 "run-in" nights followed by 12 consecutive nights after receiving placebo (14 nights/2 weeks total). No change in objective sleep duration would be demonstrated compared to baseline

SECONDARY OUTCOMES:
Change in Emotion Regulation During Melatonin Administration as Evidenced by the Emotion Regulation Index for Children and Adolescents (ERICA) | Change between baseline and two weeks
  The Emotion Regulation Index for Children and Adolescents (ERICA) is a 16-item adolescent-report measure with scores ranging from 16 to 80 (higher scores indicative of better emotion regulation). This measure will be administered during baseline and after 14 days (2 weeks) including a 2 day "run-in" followed by 12 days of melatonin administration. It is expected that emotion regulation will improve after melatonin administration compared to baseline. Normal emotion regulation varies by individual.
Change in Emotion Regulation During Placebo Administration as Evidenced by the Emotion Regulation Index for Children and Adolescents (ERICA) | Change between baseline and two weeks
  The Emotion Regulation Index for Children and Adolescents (ERICA) is a 16-item adolescent-report measure with scores ranging from 16 to 80 (higher scores indicative of better emotion regulation). This measure will be administered during baseline and after 14 days (2 weeks) including a 2 day "run-in" followed by 12 days of placebo administration. It is expected that emotion regulation will remain the same after placebo administration compared to baseline. Normal emotion regulation varies by individual.

CONTACTS AND LOCATIONS:
Overall Officials: Tori Van Dyk, PhD, Principal Investigator — Loma Linda University
Locations (2):
- United States (2):
  - Loma Linda University, Loma Linda, California
  - Loma Linda U, Loma Linda, California

IPD SHARING:
Plan to Share IPD: No